CLINICAL TRIAL: NCT02924480
Title: Intravenous Lidocaine in the Perioperative Setting and the Effects on Postoperative Pain and Bowel Function Following Cystectomy: A Pilot Study
Brief Title: Intravenous Lidocaine for Cystectomy Procedures
Acronym: Lidocaine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CAMC Health System (Other)
Responsible Party: Principal Investigator, Samuel Deem, DO, Urology Surgeon, CAMC Health System
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 16-247
Record Dates: First submitted 2016-10-03; First posted 2016-10-05 (Estimated); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Invasive Bladder Cancer
Keywords: invasive bladder cancer; cystectomy; high grade bladder cancer
MeSH Terms: interventions — Cystectomy; Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine Study Group (Active Comparator): Intravenous Lidocaine for Cystectomy Procedures: During the surgery, the lidocaine infusion group will receive the lidocaine bolus (1.5mg/kg bolus followed by a 2mg/kg/h infusion) 30 minutes prior to skin incision and the infusion will continue until 60 minutes after skin closure.
  Interventions: Procedure: Cystectomy; Drug: Lidocaine
- Placebo Study Group (Placebo Comparator): Intravenous Saline for Cystectomy Procedures: During the surgery, patients will be randomized to the control group and receive a normal saline bolus 30 minutes prior to skin incision and the infusion will continue until 60 minutes after skin closure.
  Interventions: Procedure: Cystectomy; Drug: Saline

INTERVENTIONS:
Procedure: Cystectomy
Drug: Lidocaine — Patients will receive lidocaine infusion during surgery
  Arms: Lidocaine Study Group
Drug: Saline — Patients will receive saline infusion during surgery
  Arms: Placebo Study Group

SUMMARY:
Patients scheduled for a cystectomy at Charleston Area Medical Center (CAMC) will be enrolled into a randomized, double blinded clinical trial to assess if postoperative pain and ileus are reduced by perioperative intravenous lidocaine infusion versus placebo. The hypothesis is that patients receiving the lidocaine infusion will experience better pain control and ileus resolution. It is believed that lidocaine patients will also have less opioid requirement, less mortality, a shorter length of stay, less nausea /vomiting, and fewer adverse events.

DETAILED DESCRIPTION:
Design

The design will be a randomized, double blinded, single institute prospective study with patients undergoing Open or Robotic Assisted cystectomy procedures at Charleston Area Medical Center in Charleston, West Virginia. All patients following informed consent that meet the inclusion criteria are eligible to participate in the study.

Procedures and Protocol

This study will have two groups. Each group will follow a standardized post cystectomy protocol to reduce confounding factors in regards to postoperative management.

Study Group

Group A: The lidocaine infusion group will receive the lidocaine bolus 30 minutes prior to skin incision and the infusion will continue until 60 minutes after skin closure.

Control Group

Group B: Patients will be randomized to the control group and receive a normal saline bolus and infusion in the same procedure as the study arm.

All patients in both groups will have pain scores documented at the time of the surgery. A baseline level of abdominal pain will be assessed using a 0 to 10 verbal analog scale (VAS), in which a rating of "0" indicates "no pain" and a score of "10" indicates the "worst pain imaginable". This data, which is the baseline preoperative pain score, will be used by statistician for data analysis.

After surgery, nursing staffs will record the exact time the patient passes first flatus and have first bowel movements; nurses will also routinely asked each patients of these bowel activities during the patient assessments. Postoperative nausea and/or vomiting will be assessed in a similar fashion by the nursing staff. From Postoperative Day 1 until discharge (or up to 108 hours), at specified time intervals patients will be asked to score the average pain on a scale of O-10 (0 = none; 10 = worst pain imaginable) and any nausea/vomiting was experienced. The numeric rating scale is being used in this study because it is used commonly in patients post-operatively and due to its common use in other pain assessment studies. This information along with medication use during the same time intervals will be recorded by the nursing staffs at Charleston Area Medical Center.

The American Pain Society Patient Outcome Questionnaire (APS-POQ-R) will be used to assess pain management during the first 24 hours after surgery. This questionnaire measures six aspects of pain including: pain severity and relief; impact of pain on activity, sleep, and negative emotions; side effects of treatment; helpfulness of information about pain treatment; ability to participate in pain treatment decisions; and use of nonpharmacological strategies. This has been validated in multiple studies to assess pain of patients and can be used in reference to other literature in regards to pain management previously published.

In order to compare each arm for primary outcomes, namely improved pain control, decreased opioid consumption, and improved resolution of ileus, a descriptive analysis will be performed with means, standard deviations, ranges and percentages being reported for the prospective variables. In addition subgroup analysis will be conducted using statistical tests between study and control group to examine the differences between medication use, pain relief satisfaction, and post procedure pain scores. Continuous variables will be analyzed using the Student's t-test and categorical variables using chi-square or Fisher's Exact Test. Logistic regression will be used if needed to determine if any the variables are associated with study group. A p < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing a cystectomy with an American Society of Anesthesiologists physical status classification (ASA) of 1 or 2.

Exclusion Criteria:

* Any patients with a history of substance abuse, allergy to amides, and current treatment with antiarrhythmic medications (due to lidocaine being a class 1b antiarrhythmic agent) will be excluded.
* Patients will also be excluded if they are pregnant or have a history of chronic pain syndrome, chronic bowel or liver dysfunction.
* Patients with chronic opioid use, and therefore opioid tolerance, and history of opioid addiction will also be excluded due to likely increased opioid needs for equivalent pain control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-10-12 (Actual); Primary Completion 2020-06-17 (Actual); Study Completion 2020-06-17 (Actual)

PRIMARY OUTCOMES:
Reduced pain post-operatively using verbal analog score | 108 hours after surgery
  Use verbal analog score to assess patients pain and compare between study and control groups. This will determine if patients in the lidocaine study arm experience less pain than those in the placebo group.
Time until Ileus resolution | 108 hours after surgery
  Time to ileus resolution will be compared between study and control groups using the end of surgery time to the time of first bowl movement. This should determine if those in the lidocaine study arm experience quicker Ileus resolution compared to those in the placebo study arm.

SECONDARY OUTCOMES:
Pain management during the first 24 hours after surgery using the American Pain Society Patient Outcome Questionnaire (APS-POQ-R) | 24 hours post-operatively
  The American Pain Society Patient Outcome Questionnaire (APS-POQ-R) will be used to assess pain management during the first 24 hours after surgery. This questionnaire measures six aspects of pain including: pain severity and relief; impact of pain on activity, sleep, and negative emotions; side effects of treatment; helpfulness of information about pain treatment; ability to participate in pain treatment decisions; and use of nonpharmacological strategies. These results will be compared between the lidocaine study group and the placebo study group to determine if the lidocaine study group experienced better pain management within the first 24 hours after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel G Deem, DO, Principal Investigator — CAMC Health System
Locations (1):
- Urology center of charleston, Charleston, West Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided